CLINICAL TRIAL: NCT01325675
Title: Aerobic Interval Training in Patients With Paroxysmal or Persistent Atrial Fibrillation
Brief Title: Aerobic Interval Training in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2010/3345-1(REK)
Record Dates: First submitted 2011-03-23; First posted 2011-03-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Motor activity
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval training (Experimental): Interval training
  Interventions: Behavioral: Interval training
- Control (No Intervention): Live as usual

INTERVENTIONS:
Behavioral: Interval training — Aerobic interval training will be performed with 4 times of 4 minutes intervals at an intensity of 90-95% of maximum heart rate and active pauses of 3 minutes between intervals. 3 times a week for 12 weeks.
  Arms: Interval training

SUMMARY:
The purpose of this study is to determine the effect of aerobic interval training in patients with paroxysmal or persistent atrial fibrillation, especially to see if the burden of atrial fibrillation and symptoms are reduced.

DETAILED DESCRIPTION:
Long term endurance sport practice is associated with a higher incidence of atrial fibrillation. Moderate/light physical activity seems to be associated with a lower incidence. The underlying mechanisms are uncertain. In order to examine the effect of training in this population, the investigators will perform a randomised controlled study with aerobic interval training in patients with paroxysmal/persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent atrial fibrillation, that are able to perform aerobic interval training.

Exclusion Criteria:

* Performing high intensity training (pulse >90% of max) for more than 2 times a week.
* Moderate intensity training more than 30 min, more than 3 times a week
* Previous open heart surgery
* EF <40%
* Significant aorta stenosis
* Mitral insufficiency, >gr. 2
* Pacemaker
* Earlier coronary intervention and not complete revascularization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in burden of atrial fibrillation | Baseline and 4 weeks after ended intervention period
  Burden of atrial fibrillation(number of episodes, duration(percent of the day)) continually measured, and reported by the patient. Analysed for the patients in total, with sub analysis in the groups of paroxysmal and persistent AF and in those with a low burden of atrial fibrillation vs. those with a larger burden.

SECONDARY OUTCOMES:
Size of left atrium and ventricle | Baseline and after ended intervention period(12 weeks)
  Atrial and ventricular size will be evaluated by echocardiography and MRI.
Blood samples | Baseline and after ended intervention period(12 weeks)
  Interleukin-6, pro-BNP, d-dimer and von Willenbrands factor are measured.
Endothelial function | Baseline and after ended intervention period(12 weeks)
  FMD
Atrial extrasystoles | Baseline and after ended intervention period(12 weeks)
  Atrial extrasystoles on 48h Holter monitoring. Will alse be measured in the first week of training.
Ablation procedure | Measured during the ablation procedure (day 1)
  Duration of ablation, number of ablation points, success.
Maximal oxygen uptake | Baseline and after ended intervention period(12 weeks)
Atrial and ventricular function | Baseline and after ended intervention period(12 weeks)
  Atrial and ventricular function measured by MR and echocardiography
Fibrosis | Baseline and after ended intervention period(12 weeks)
  Fibrosis in left atrium and left ventricle measured by MRI.
Quality of life | Baseline and after ended intervention period(12 weeks)
  Measured with SF-36, Symptom and Severity Checklist and EHRA score of AF- related symptoms
Burden of atrial fibrillation in the intervention period | Week 1-4, 5-8 and 9-12
  The intervention period is divided into 3 periods of 4 weeks each. The mean burden of atrial fibrillation(percent of time with atrial fibrillation) and number of episodes in each of those periods will be assessed to see if exercise changes the amount of fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paal Loennechen, PhD, Study Chair — St. Olavs Hospital; Ulrik Wisløff, PhD, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Malmo V, Nes BM, Amundsen BH, Tjonna AE, Stoylen A, Rossvoll O, Wisloff U, Loennechen JP. Aerobic Interval Training Reduces the Burden of Atrial Fibrillation in the Short Term: A Randomized Trial. Circulation. 2016 Feb 2;133(5):466-73. doi: 10.1161/CIRCULATIONAHA.115.018220. Epub 2016 Jan 5. PMID 26733609